CLINICAL TRIAL: NCT01238003
Title: Clinical Relevance of Anti-Neutrophil Cytoplasm Antibody (ANCA)in Hospitalized Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Nina Avshovich, Hillel Yaffe Medical Center
Other Study IDs: HYMC-10-0087
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: ANCA-related Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hospitalized patients
  Interventions: Other: Interpretation of blood test results

INTERVENTIONS:
Other: Interpretation of blood test results — Interpretation of blood test results

SUMMARY:
Laboratory testing of Anti-Neutrophil Cytoplasm Antibody (ANCA) is used to confirm diagnosis of patients who have a high level of suspicion for ANCA-related vasculitis. In these patients the specificity and sensitivity to the ANCA test is very high. This study hopes to prove that when this lab test is performed on blood of patients who do not have a high level of suspicion for ANCA-related vasculitis, the sensitivity and specificity is reduced and there are many false positive results. Because of this, it should not be used as a screening test for a more general patient population.

ELIGIBILITY:
Inclusion Criteria:

* Blood samples sent for ANCA lab test

Exclusion Criteria:

* Patients with ANCA vasculitis
* Patients with known malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in internal medicine ward
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Mostly negative lab results | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel